CLINICAL TRIAL: NCT00004033
Title: Phase II Clinical Study of a Liposome Entrapped Cisplatin Analog (L-NDDP) Administered Intrapleurally in Patients With Malignant Pleural Mesothelioma
Brief Title: Liposomal-Cisplatin Analogue (L-NDDP) in Treating Patients With Malignant Pleural Mesothelioma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000066141; P30CA016087 (NIH); NYU-9850; MDA-FDR001234; MDA-ID-95209; NCI-G99-1575
Record Dates: First submitted 1999-12-10; First posted 2004-04-15 (Estimated); Last update posted 2011-03-28 (Estimated); Status verified 2011-03

CONDITIONS: Malignant Mesothelioma
Keywords: localized malignant mesothelioma; advanced malignant mesothelioma; recurrent malignant mesothelioma
MeSH Terms: conditions — Mesothelioma, Malignant | interventions — bis-neodecanoato-1,2-diaminocyclohexaneplatinum(II)

INTERVENTIONS:
Drug: liposomal NDDP
Procedure: therapeutic thoracoscopy

SUMMARY:
RATIONALE: Patient abstract not available

PURPOSE: Patient abstract not available

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the antitumor efficacy of a liposomal-cisplatin analogue (L-NDDP) administered into the pleural space in patients with malignant pleural mesothelioma. II. Determine the time to progression and overall survival in this patient population. III. Evaluate the quantitative and qualitative toxicity of intrapleural L-NDDP.

OUTLINE: All patients undergo a thoracoscopy under general anesthesia. The thoracoscope is removed and any collected fluid is drained from the chest cavity. The first treatment with liposomal-cisplatin analogue (L-NDDP) is administered at this time into the intrapleural space over a 10 minute period. Subsequent 10 minute intrapleural infusions of L-NDDP through a percutaneous catheter are administered every 3 weeks. Treatment continues unless unacceptable toxic effects or disease progression occurs. Antitumor activity is assessed 2 months after the second course of therapy, and every 2 months thereafter.

PROJECTED ACCRUAL: A total of 14-30 patients will be accrued for this study within 2.5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Pathologically confirmed malignant pleural mesothelioma Free flowing pleural effusion

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: Zubrod 0-2 Life expectancy: At least 12 weeks Hematopoietic: WBC greater than 4,000/mm3 Granulocyte count greater than 1,500/mm3 Platelet count greater than 100,000/mm3 Hepatic: Bilirubin no greater than 1.5 mg/dL SGPT no greater than 1.5 times upper limit of normal Renal: Creatinine no greater than 1.5 mg/dL Cardiovascular: No unstable angina No clinical evidence of congestive heart failure Pulmonary: No postobstructive pneumonia Other: Fertile patients must use effective contraception Not pregnant or nursing No serious concurrent infection No prior malignancies except basal cell or squamous cell skin carcinomas, stage I colon, cervical, breast, prostate, head and neck, or lung cancer, as long as there has been no evidence of tumor occurrence within the past 5 years

PRIOR CONCURRENT THERAPY: Biologic therapy: At least 3 weeks since prior biologic therapy No concurrent immunotherapy Chemotherapy: No prior chemotherapy No concurrent chemotherapy Endocrine therapy: At least 3 weeks since prior hormonal therapy No concurrent hormonal therapy Radiotherapy: No prior chest radiotherapy At least 3 weeks since other prior radiotherapy No concurrent radiotherapy Surgery: Prior pleurodesis or chest surgery on the same side of the effusion is allowed as long as there is a free flowing pleural effusion without loculation At least 2 weeks since major surgery other than biopsy Other: At least 3 weeks since use of any other investigational medication No concurrent use of any other investigational medications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 1998-09; Primary Completion 2001-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Abraham Chachoua, MD, Study Chair — NYU Langone Health
Locations (2):
- United States (2):
  - NYU School of Medicine's Kaplan Comprehensive Cancer Center, New York, New York
  - University of Texas - MD Anderson Cancer Center, Houston, Texas